CLINICAL TRIAL: NCT02823613
Title: The Influence of High and Low Salt on Exosomes in the Urine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Diabetes Academy (Other); Odense University Hospital (Other); Beckett Foundation (Other)
Responsible Party: Principal Investigator, Rikke Zachar Langkilde, MD, phd student, University of Southern Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RZL-SDU-IMM-CVR
Record Dates: First submitted 2016-06-23; First posted 2016-07-06 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: ENaC; Exosomes; Urinary biomarker; Salt regulation

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy male test subjects 1-5 (Experimental): High salt diet followed by low salt diet
  Interventions: Dietary Supplement: High salt diet followed by low salt diet
- Healthy male test subjects 6-10 (Experimental): Low salt diet followed by high salt diet
  Interventions: Dietary Supplement: Low salt diet followed by high salt diet

INTERVENTIONS:
Dietary Supplement: High salt diet followed by low salt diet — High salt diet (250 mmol/day) in 5 days followed by low salt diet (60-70 mmol/day) in 5 days.
  Arms: Healthy male test subjects 1-5
Dietary Supplement: Low salt diet followed by high salt diet — Low salt diet (60-70 mmol/day) in 5 days followed by high salt diet (250 mmol/day) in 5 days.
  Arms: Healthy male test subjects 6-10

SUMMARY:
The hypothesis is that changes in the epithelial sodium channel (ENaC) in the kidney is reflected in urinary exosomes and that the amount of ENaC as well as the cleavage degree is upregulated in conditions with low salt.

DETAILED DESCRIPTION:
Methods:

Exosomes will be isolated from spot urine by ultracentrifugation and tested using western blotting. In-house developed antibodies against different parts of the ENaC gamma subunit as well as commercial antibodies will be used. A marker for exosomes will validate the presence of exosomes in the urine.

Power considerations:

In this cross over salt-intervention study with quantification of ENaC the investigators refer to a published study regarding the sodium-chloride co-transporter (NCC) in the kidney, were rats where given aldosterone infusion or a low salt diet. In this study n=6 was sufficient to detect a 2-3 fold change in NCC in urinary exosomes. Furthermore 5 patients with primary aldosteronism had a significant increase in NCC in urinary exosomes (N. Lubbe et al, Hypertension 2012).

On the basis of this the investigators choose to test 10 persons, but are not able to make a regular power calculation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 20-40
* Body Mass Index (BMI, weight/height^2) between 18 and 25.

Exclusion Criteria:

* Increased blood pressure (hypertension) or in treatment for high blood pressure
* Diabetes
* Regular medical intake
* Smoking
* Expectation of lacking cooperation or lack of understanding of the experiment
* Clinical relevant organic or systemic disease including malign disease
* Decreased kidney function

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Changes in epithelial sodium channel (ENaC) appearance in urinary exosomes | After 5 days on high or low salt diet
  Semiquantitative western blotting

SECONDARY OUTCOMES:
Plasma aldosterone | Before study start and after 5 days on high or low salt diet
  Concentration in plasma.
Renin | Before study start and after 5 days on high or low salt diet
  Concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Boye L Jensen, dr.med., phd, Study Director — Cardiovascular and Renal Research, Institute of Moleculare Medicine, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zachar RM, Skjodt K, Marcussen N, Walter S, Toft A, Nielsen MR, Jensen BL, Svenningsen P. The epithelial sodium channel gamma-subunit is processed proteolytically in human kidney. J Am Soc Nephrol. 2015 Jan;26(1):95-106. doi: 10.1681/ASN.2013111173. Epub 2014 Jul 24. PMID 25060057
- [Background] van der Lubbe N, Jansen PM, Salih M, Fenton RA, van den Meiracker AH, Danser AH, Zietse R, Hoorn EJ. The phosphorylated sodium chloride cotransporter in urinary exosomes is superior to prostasin as a marker for aldosteronism. Hypertension. 2012 Sep;60(3):741-8. doi: 10.1161/HYPERTENSIONAHA.112.198135. Epub 2012 Jul 30. PMID 22851731